CLINICAL TRIAL: NCT04825782
Title: A Pregnancy Registry to Assess the Safety of Antimalarial Use in Pregnancy
Brief Title: MiMBa Pregnancy Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Medicines for Malaria Venture (Other); Worldwide Antimalarial Resistance Network (Network); Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20-056
Record Dates: First submitted 2021-02-23; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Malaria in Pregnancy; Pregnancy Related; Congenital Anomaly
Keywords: Malaria; Pharmacovigilance; Pregnancy registry; Antimalarials
MeSH Terms: conditions — Congenital Abnormalities; Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Women exposed to antimalarials during pregnancy: Pregnant women will be followed up prospectively. In certain sites, women of childbearing age (15-49 years) will be enrolled prior to pregnancy to ensure early pregnancy detection. Pregnancy and infant outcomes will be assessed systematically and recorded.
- Pregnant Women unexposed to antimalarials during pregnancy: Pregnant women will be followed up prospectively. In certain sites, women of childbearing age (15-49 years) will be enrolled prior to pregnancy to ensure early pregnancy detection. Pregnancy and infant outcomes will be assessed systematically and recorded.

SUMMARY:
The MiMBa (Malaria in Mothers and Babies) Pregnancy Registry aims to generate robust evidence on the safety of a range of antimalarials when used in pregnancy, particularly in the first trimester. This will be a multi-country observational study and will be deployed in several field sites in Africa.

DETAILED DESCRIPTION:
Background:There is often no, or limited, safety data on drug use in early pregnancy and particularly for drugs targeting tropical diseases because these are not widely used in resource-rich countries with robust pharmacovigilance systems. It is critical to develop surveillance systems to assess the safety of these drugs in pregnancy. Malaria in pregnancy requires prompt and effective treatment to prevent adverse health consequences for the mother and her unborn baby. Malaria infection in the first trimester has been associated with miscarriage, preterm birth and low birth weight. Pregnant women in the first trimester are often inadvertently treated with the same antimalarials as provided to the adult population which is a concern for drugs which are contraindicated in early pregnancy, such as artemisinin combination therapies (ACTs). This occurs either because they are not aware or do not report that they are pregnant, or because quinine, the standard of care for malaria treatment in the first trimester is not available. There is limited data available about the safety of ACTs in early pregnancy. Investigators will develop a pregnancy registry for monitoring the safety of antimalarial drugs during pregnancy with a focus on the first trimester.

Overall Aim: The aim of the pregnancy registry is to generate robust data on the safety of a range of antimalarials in pregnancy and particularly use in the first trimester to inform regulators and policymakers.

Methods in Brief: Investigators will set-up a pregnancy exposure registry for antimalarial drugs to capture safety data from women inadvertently exposed to (i.e. treated with) antimalarials used in the general population that are not currently recommended for use in the first trimester. To capture this safety data, several sentinel sites will be set-up in multiple malaria-endemic countries to follow women from the moment the pregnancy is identified and capture pregnancy outcomes (i.e. miscarriage, stillbirth, live birth). Some sites (including Kenya) will provide pregnancy tests to enable early pregnancy detection and referral to ANC to capture early miscarriages. Newborns will be assessed for congenital anomalies at birth and up to 2 years of age. Any suspected case of congenital anomalies will be referred for further assessment by a specialist (e.g. paediatrician) who will confirm the diagnosis and advise on how to further manage any problems or complications. The national referral system will be used in cases requiring further intervention. Exposure data will be collected on any acute illnesses occurring during pregnancy, such as malaria and COVID-19, and chronic conditions, such as HIV, TB, epilepsy or diabetes, and details of any treatment given (including antimalarials). Antimalarial and other drug exposure data in early pregnancy, i.e. before the pregnancy was known, will be captured through record linkage with treatment records from outpatient departments, community health workers, and any other treatment records. Women will provide informed consent for this data to be collected and to be followed up throughout pregnancy. The pregnancy outcomes and prevalence of congenital anomalies will then be compared between pregnancies exposed and those not exposed to specific antimalarials during the first trimester.

Expected Outcomes: The expected outcome of this study is information and reassurance about the safety profile of specific antimalarials, with a focus on the first trimester, to inform malaria treatment guidelines. The findings will be shared with the relevant local and national health and regulatory authorities and disseminated in scientific meetings and in peer-reviewed journals. Data generated will be pooled with data from similar pregnancy registries in other malaria-endemic countries and will be shared with the WHO/TDR Central registry for epidemiological surveillance of drug safety in pregnancy and other relevant pregnancy exposure registries.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or women of childbearing age (15-49 years)

  * Resident within the defined catchment area. Residency status will be defined as having resided in the area for at least four months.
  * Willingness to attend antenatal care and deliver in the study area.
  * Willingness to give informed consent (and assent for non-pregnant WOCBAs under 18 years of age).

Exclusion Criteria:

* Refusal to participate or be followed up to the end of pregnancy. • Any medical, psychiatric, or social condition that would interfere with the ability to provide an accurate medical or drug history or the volunteer's ability to give informed consent (e.g. mentally disabled patients).

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women
Study Population: Women of childbearing age (40,000 to 60,000) and Pregnant Women - approximately 3000 to 5500 per year
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Miscarriage | Between pregnancy identification and 28 weeks gestation
  Spontaneous pregnancy loss <28 weeks gestation
Stillbirth | Between pregnancy identification and delivery
  A confirmed pregnancy lasting until 28 weeks of pregnancy, that results in the birth of a baby showing no signs of life
Major congenital anomalies | Up to 12 months after birth
  Structural abnormality with surgical, medical or cosmetic importance that is present at birth

SECONDARY OUTCOMES:
Maternal Mortality | Up to 6 weeks post-delivery
  Maternal mortality up to 6 weeks post-delivery
Neonatal mortality | By 28 days post-delivery
  Infant death by ≤28 days of birth
Low birthweight | Within 48 hours of birth
  Birth weight<2500gr
Prematurity | At delivery
  Delivery ≤37 completed weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Feiko ter Kuile, MD, PhD, Study Director — Liverpool School of Tropical Medicine
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
The full anonymised research database will be made publicly available as soon as the full study findings have been published or based on any data requests that may occur during the study or analysis is still ongoing. For the databases, we will use a controlled access approach. The data sharing policy will be provided in publications and on the respective websites.